CLINICAL TRIAL: NCT05607732
Title: Primary Care Detection of Cognitive Impairment Leveraging Health & Consumer Technologies in Underserved Communities: The MyCog Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Oak Street Health (Unknown); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: U01NS105562 (NIH)
Record Dates: First submitted 2022-11-02; First posted 2022-11-07 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Cognitive Impairment; Cognitive Decline; Alzheimer Disease
Keywords: Detect; Manage
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyCog Paradigm (Experimental): The MyCog paradigm establishes a protocol for implementing our self-administered assessment in the clinic whenever a patient or involved family member reports a concern. The MyCog test can be completed either in the exam room or the waiting room. The MyCog app, on an iPad, can be readily linked to the electronic health record, so once the two tests are completed, results are securely transmitted and will populate within discrete, fields that can be queried found in the patient record; specifically: 1) in a screening tab, under 'cognitive abilities', 2) a flow sheet to capture trend with future repeated tests - informing physicians of a patient's relative vs. normative cognitive decline. Both a binary, objective classification of 'impairment detected or suspected' or 'no impairment detected' will populate in the record, as well as a summary score to further guide the clinician by clarifying the extent to which a patient's performance falls outside a normal threshold.
  Interventions: Diagnostic Test: MyCog
- Usual Care Arm (No Intervention): At Oak Street Health, cognitive assessments included when concerns are reported by patients or family members, if a clinician suspects a concern, or during Annual Wellness Visits (AWVs) are limited to the Mini-Cog©, and are variably administered, particularly outside of AWVs. Oak Street practices vary by clinician in terms of making referrals, how results are documented, what diagnosis code, placement in problem list or visit diagnosis, and any follow-up plans. While we will not make any explicit recommendations to usual care practices regarding their use of a cognitive assessment, we will ensure that 1) any chosen test is linked to a data field that can be queried in the EHR, and 2) providers receive a compiled list of local medical and non-medical referrals for any detected cases of CI. The Alzheimer's Association recommendations for early detection efforts among primary care practices will be provided to each clinical leadership.

INTERVENTIONS:
Diagnostic Test: MyCog — MyCog uses well-validated, self-administered, iPad-based measures from the NIH Toolbox for the Assessment of Neurological Behavior and Function Cognition Battery to provide an efficient and sensitive cognitive screen that can be easily implemented in primary care. Preliminary data shows these tests can discriminate between cognitively normal older adults and those with CI (specifically mild cognitive impairment); enabling physicians to assess CI in ways currently not available.
  Arms: MyCog Paradigm

SUMMARY:
Our study intends to offer 'real world' evidence of a viable, sustainable means to mobilize primary care via a comprehensive strategy for detecting cognitive impairment and dementias, advancing next steps for referral, and participating in the care planning and management of affected patients and caregivers. We will conduct a clinic-randomized, pragmatic trial testing the effectiveness and fidelity of our NIH Toolbox-derived paradigm to improve early detection and management of cognitive impairment/dementia in primary care settings serving health disparate patient populations.

DETAILED DESCRIPTION:
Practical, scalable strategies are needed to help primary care practices better detect and manage cognitive impairment (CI), especially those caring for medically underserved, low socioeconomic status (SES) communities. Since 2017, our team has been a member of the Consortium for Detecting Cognitive Impairment, Including Dementia (DetectCID); a network dedicated to improving clinical paradigms for early detection of CI and Alzheimer's disease-related dementias (ADRD) and its subsequent management in everyday clinical settings. Having developed the NIH Toolbox for Assessment of Neurological and Behavioral Function and with expertise in health system re-design for patient-centered care, we validated our clinical paradigm, known as MyCog. This includes a brief, iPad-based, self-administered, electronic health record (EHR)-linked strategy to assess for CI during primary care visits when concerns are identified, and 'turnkey' recommendations to address them.

We will partner with a national primary care provider (Oak Street Health) and conduct a 2-arm, clinic-randomized, 'real world' pragmatic trial comparing MyCog to usual care. We will focus on populations experiencing CI/ADRD disparities: Black, H/L, and low SES older adults.

Our specific aims and hypotheses (H) are to:

Aim 1: Test the effectiveness of the MyCog paradigm to improve early detection of cognitive impairment and dementias among low SES, Black and Hispanic/Latino older adults.

Compared to usual care, primary care practices implementing MyCog will demonstrate:

H1: higher rates of detected and/or diagnosed cases of cognitive decline and impairment

Among detected and/or diagnosed cases of cognitive impairment, primary care practices implementing MyCog - compared to usual care - will have:

H2: a greater proportion of early stage (mild) cognitive impairments H3: more referrals for related medical and non-medical services H4: greater caregiver involvement in subsequent patient visits

Aim 2: Investigate the presence of disparities in early detection of cognitive impairment, its diagnosis, and rate of referrals by race and ethnicity.

H5: Disparities in early detection of CI, diagnosis, and referrals by race and ethnicity will be reduced among those primary care practices implementing MyCog compared to usual care.

Aim 3: Determine the fidelity and reliability of MyCog and identify any patient, caregiver, clinician, and/or health system barriers to its optimal, sustained implementation.

Aim 4: Assess the cost-effectiveness of the MyCog paradigm from a primary care perspective.

ELIGIBILITY:
Inclusion Criteria:

* been seen by an Oak Street healthcare provider affiliated with one of the 24 enrolled practices
* had at least one clinic visit (routine or Annual Wellness Visit) during the 3-year study period
* not been diagnosed previously with cognitive deficits, impairments or dementias.

Exclusion Criteria:

* Children, adolescence, and younger adults are excluded as cognitive impairment in these populations is often due to differences other than age-related changes.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45257 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
Rate of detected impairment | 3 years
  This will be operationalized as either results of an administered cognitive test suggesting impairment ('detected') or having any relevant International Classification of Diseases (ICD) 10 code recorded in a patient's record after the trial launch date and throughout follow-up observation period ('diagnosis').

SECONDARY OUTCOMES:
Rate of detected cases with mild impairment | 3 years
  Mild vs. other impairment rates will be compared across trial arms, operationalized by ICD code groupings.
Rate of cognition-related referrals | 3 years
  Extraction from the electronic data warehouse for whether or not a cognitive-related referral was made (medical or non-medical) following a "detected" cognitive screen
Caregiver Involvement | 3 years
  Text search of clinic note from any follow-up visit post AWV, wellness visit mention of accompanying family member/caregiver; extraction from Enterprise Data Warehouse to determine if proxy access to patient's MyChart portal has been shared.

CONTACTS AND LOCATIONS:
Locations (1):
- Oak Street Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lovett R, Bonham M, Yoshino Benavente J, Hosseinian Z, Byrne GJ, Varela Diaz M, Bass M, Yao L, Adin-Cristian A, Batio S, Kim M, Sluis A, Moran M, Buchanan DR, Hunt J, Young SR, Gershon R, Nowinski C, Wolf M. Primary care detection of cognitive impairment leveraging health and consumer technologies in underserved US communities: protocol for a pragmatic randomised controlled trial of the MyCog paradigm. BMJ Open. 2023 Oct 18;13(10):e080101. doi: 10.1136/bmjopen-2023-080101. PMID 37852774